CLINICAL TRIAL: NCT00002094
Title: Prospective Open-Label Study of the Emergence of Drug Resistance in Patients Infected With HIV-1 Who Are Taking Oral U-87201E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 117A; M/3330/0007
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-02

CONDITIONS: HIV Infections
Keywords: Virus Replication; Acquired Immunodeficiency Syndrome; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — atevirdine

INTERVENTIONS:
Drug: Atevirdine mesylate

SUMMARY:
To determine the time course of development of resistance to atevirdine mesylate ( U-87201E ) in patients with HIV isolates showing in vitro resistance to zidovudine ( AZT ). To determine the genotype changes in HIV reverse transcriptase associated with in vitro AZT resistance to U-87201E. To determine the genotype and phenotype effects of treatment with a nondideoxynucleoside agent on the alterations of the HIV-1 population associated with in vitro AZT resistance. To determine whether serial passage of patient pre-drug HIV isolates in the presence of U-87201E will generate the resistant mutants that may subsequently emerge in the patients.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Enrollment on protocol RV-43 (AZT resistance study).
* Development of a primary RV-43 study endpoint-opportunistic infection.
* HIV isolate with an AZT IC50 > 50 times that of the sensitive type strain.
* Able to swallow tablets without difficulty.
* Normal QTc interval on EKG.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Clinically significant hypersensitivity to piperazine type drugs (Antepar, Stelazine).
* Severe uncontrollable diarrhea or vomiting or known malabsorption.
* Symptomatic hyperlipidemia.

Concurrent Medication:

Excluded:

* Other experimental drugs.
* AZT, ddI, ddC, foscarnet, immunomodulators or other agents with primary antiretroviral activity (exemptions by principal investigator permitted).

Patients with the following prior conditions are excluded:

History of clinically significant cardiovascular disease or nervous system or muscle disease, including seizures, peripheral neuropathy, dementia, or motor dysfunction.

Prior Medication:

Excluded:

* Experimental drugs within 4 weeks prior to study entry.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Natl Naval Med Ctr, Bethesda, Maryland, United States